CLINICAL TRIAL: NCT03680456
Title: Postoperative Replacement of Intraoperative Iron Losses
Acronym: POREIIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kepler University Hospital (Other)
Responsible Party: Principal Investigator, Roxane Brooks, Principal Investigator, Kepler University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPL107
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Blood Loss Anemia
Keywords: Anemia; Ferric carboxymaltose; intravenous iron; intraoperative blood loss; patient blood management; Red blood cell transfusion; postoperative iron replacement
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; Crystalloid Solutions; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: interventional randomized doubleblind, Placebo controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): due to postoperative Hemoglobin Level intravenous iron Ferriccarboxymaltose is Infuses, dosage is based on the Ganzoni-Algorithm
  Interventions: Drug: Ferric carboxymaltose
- Placebo (Placebo Comparator): Natriumchlorid is the placebo
  Interventions: Drug: Crystalloid

INTERVENTIONS:
Drug: Ferric carboxymaltose — maximum of 750mg in U.S. is given, maximum of 1000mg in EU
  Other Names: Ferinject
  Arms: Intervention
Drug: Crystalloid — an equivalent volume dose of Natriumchlorid is administered
  Other Names: Natriumchlorid
  Arms: Placebo

SUMMARY:
By performing a randomized, blinded placebo controlled exploratory trial we speculate that replacement of perioperative, bleeding-induced iron losses with ferric carboxymaltose immediately after the surgical procedure can replenish iron with increased hemoglobin levels and reduce the amount of pRBCs transfused in the postoperative period (30 days post surgery).

DETAILED DESCRIPTION:
In the last few years, state of the art Patient Blood Management (PBM programs have been gaining worldwide attention. This may be attributed to the significant improvements in patient outcomes that follow adequate preoperative preparation and intraoperative optimization of the circulating red cell mass.

The first pillar of PBM (pre-, intra-, and postoperative optimization of red cell mass by means other than red cell transfusions including intravenous iron and erythropoietin stimulating agents) can meet significant barriers and might be difficult to implement. In daily clinical practice, timely identification and treatment of preoperative anemia is difficult to organize due to structural and behavioral constraints. Therefore, today, there are still a striking number of patients who are admitted for surgery without adequate preoperative treatment of anemia regardless of its causes. Notably, even for this patient population, it has been demonstrated by experimental and larger observational data that postoperative application of intravenous iron could help to reduce perioperative transfusions by restoring red cell mass. The complete potential of perioperative intravenous iron therapy has yet to identified, including improvements such as early mobility and other improved outcomes. Furthermore, a substantial number of patients are not included in preoperative red cell mass optimization, since the preoperative hemoglobin concentration is either high enough in terms of the thresholds of the World Health Organization (♂ 13 g/dl and ♀ 12 g/dl), or borderline (mild) anemia is diagnosed and no treatment is offered. These patients may be prone to substantial intraoperative blood losses, and as a consequence might suffer from postoperative iron restricted anemia. In fact, there are a remarkable number of patients that have adequate hemoglobin concentrations preoperatively, but ultimately develop anemia with iron deficiency postoperatively due to significant intraoperative bleeding. Data from ICU patients' with postoperative iron deficiency has significant impact on outcome including postoperative fatigue, and consequently a prolonged healing process.

Although this problem is common, current PBM strategies are in need of validation of one of the PBM guidelines: postoperative replacement of blood loss with resultant iron losses in patients without preoperative anemia thus avoiding exposure to allogeneic transfusions in this population. The untested hypothesis is that this approach could improve postoperative outcomes including mobilization. Based on a recent publication one might surmise that it is not (only) postoperative anemia, but rather untreated iron deficiency, that is responsible for a delay in postoperative mobilization and recovery. It is therefore the aim of the proposal presented to describe an additional approach, in which perioperative, surgical blood loss iron losses are replaced immediately following the surgical procedure in patients that did not receive iron preoperatively due to normal or minor reduction in hemoglobin concentrations (red cell mass). This replacement may take place in either the postoperative anesthesia care unit or in the ICU, Although preoperative treatment of iron deficiency anemia is widely considered the most important domain of perioperative iron therapy, the additional post-operative replacement is as useful as preoperative preparation and seems to be more convenient to implement.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing non-emergency

  - cardiac surgery - obstetric surgery - intra-abdominal surgery
* preoperative Hb (during the premedication visit):

  * ♂: Hb>12.5g/dl
  * ♀: Hb>11.5g/dl
* postoperative Hb (immediately after surgical procedure in the recovery room):

  - 2 g/dl below preoperative Hb concentration
* age ≥ 18 years
* Admission to intensive care unit or post-anesthesia care unit
* Able to sign consent for the trial

Exclusion Criteria:

* age < 18 years
* emergency surgery
* perioperative application of iron and/or erythropoietin
* intraoperative transfusion of allogeneic erythrocytes
* known hemochromatosis
* known allergic reaction linked to iron medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Hemoglobin Level | 30days
  Hemoglobin in g/dl

SECONDARY OUTCOMES:
Number of RBCs | 30days
  Number of Units of Red Blood Cell transfusions
10 Feet Walking test | day 7 and 30 post randomization
  ability to walk 10 feet or across the room
6min Walking Test | preoperative day, day 7 and 30
  The distance ist measured which the Patient is able to walk in 6 min
Infection | 30 Days
  Number of severe Sepsis or wound infection due to SSC Guidelines and Sofa-Score
MI | 30days
  myocardial infarction is diagnosed du to ECG, Troponin T and clinical signs and symptoms for myocardial infarction e.g. chest pain
AKI | 30 days
  acute kidney injury due to KDIGO criteria
Stroke | 30days
  numbers of stroke (e.b. subarachnoid hemorrhage and others)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Meier, Prof, Study Director — Kepler University Hospital, JKU Linz
Locations (1):
- Universitätsklinik für Anästhesie und Intensivmedizin, Linz, Austria

IPD SHARING:
Plan to Share IPD: No